CLINICAL TRIAL: NCT03066128
Title: Point-of-care Viral Load Testing to Enable Streamlined Care and Task Shifting for Chronic HIV Care
Acronym: STREAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Paul Drain, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00001466; R21AI124719 (NIH)
Record Dates: First submitted 2017-02-22; First posted 2017-02-28 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Chronic HIV Infection
Keywords: Task shifting; HIV care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the Intervention Group will receive chronic ART management from a Professional Nurse and/or Enrolled Nurse every 2 months, and if stable after 6 months, community pharmacy ART collection through CCMDD. Viral load monitoring will be by a point-of-care viral load testing.
  Interventions: Diagnostic Test: Point-of-care viral load testing
- Standard of Care (Experimental): Participants in the Standard-of-Care control arm will receive the standard-of-care for the clinic consisting of visits with a professional clinician (Physician or Professional Nurse) and once stable, community pharmacy ART collection through CCMDD.Viral load monitoring will be by lab-based viral load testing
  Interventions: Other: Lab-based viral load testing

INTERVENTIONS:
Diagnostic Test: Point-of-care viral load testing — Point-of-care viral load testing will be performed while the participant is in the clinic to ensure that participants receive the viral load results on the same day
  Arms: Intervention
Other: Lab-based viral load testing — Viral load testing will be lab based and follow standard of care procedures
  Arms: Standard of Care

SUMMARY:
Effective management of patients on antiretroviral therapy (ART) is essential to improve clinical outcomes and prevent HIV transmission, but monitoring life-long ART for over 15 million HIV-infected people has become a challenge, particularly in low- and middle-income countries (LMICs). As programs continue to focus on identifying HIV-infected people and starting ART at higher CD4 thresholds, HIV providers have been overburdened, which has resulted in falling retention rates. As ART coverage scales up to include millions more people, additional strain will be placed on HIV clinicians and laboratories to manage stable patients on chronic ART. Implementing point-of-care HIV VL testing to enable task shifting to nurses for chronic HIV care may help mitigate these burdens. Point-of-care Viral Load (VL) testing is intended to differentiate patients who are potentially failing on their ART, so that they can be referred to the next level of care for possible ART regiment change, from patients who are virally suppressed on ART and can be managed by nurses. The investigator's scientific objective is to test the clinical equivalence and reduced cost of implementing a model for chronic HIV care that uses a point-of-care HIV VL assay to enable streamlined care and task shifting among healthcare workers at an urban clinic in South Africa. The central hypothesis is that rapid HIV VL testing, implemented by nurses, is an effective and cost-efficient strategy for management of chronic HIV infection in the majority of patients, thereby allowing more resources to be directed at the minority of patients who need greater attention. This work is innovative because it uses a randomized evaluation of an implementation model that combines a novel diagnostic point-of-care test with streamlined care and task shifting among healthcare workers compared to standard of care for chronic HIV care in a resource-limited setting. This randomized trial will then form the basis of a larger, multicountry proposal to demonstrate the clinical equivalence and cost-effectiveness of implementing an integrated point-of-care HIV VL testing and streamlined care model for chronic HIV care in LMICs. If nurses using clinic-based HIV VL testing are cost-effective for achieving both viral suppression and retention in care among patients on ART, then implementation of this chronic HIV care model would alleviate the strain on existing HIV providers and laboratories in LMICs.

DETAILED DESCRIPTION:
The study design will be an open-label, randomized, non-inferiority implementation trial with 2 study arms. Patients will be enrolled when due their 6 month VL since initiating ART.

Standard of Care Arm:

Participants in the Standard-of-Care (SOC) control arm will receive the standard-of-care for the clinic consisting of visits with a professional clinician (Physician or Professional Nurse) and once stable, community pharmacy ART collection through CCMDD. Viral load monitoring will be lab-based. Participants will be assessed for clinical symptoms/signs of tuberculosis, other opportunistic infections, and ART side effects at each clinical encounter. Participants who have a high lab-based HIV VL (≥1,000 copies/mL) will receive intensive adherence counseling and be asked to return to the clinic in 2 months for repeat HIV VL testing. If the HIV VL remains high (≥1,000 copies/mL) after the 2 months of intensive adherence counseling, then the patient will be switched to a second-line ART regimen by a physician.

Intervention Arm:

Participants in the Intervention Group will receive chronic ART management from a Professional Nurse and/or Enrolled Nurse every 2 months, and if stable after 6 months, community pharmacy ART collection through CCMDD. Viral load monitoring will be POC. Enrolled Nurse visits will consist of a clinical symptom and ART side effect checklists, and an ART adherence questionnaire, which trigger up-referral to a Professional Nurse/MO where appropriate. Point-of-care Xpert® HIV-1 VL testing will be performed while the participant is in the clinic to ensure that participants receive the VL results on the same day. Participants who have a high HIV VL (≥1,000 copies/mL) will be referred to a Professional Nurse. As with the standard-of-care arm, they will receive intensive adherence counseling and be asked to return to the clinic in 2 months for repeat point-of-care Xpert® HIV-1 VL testing. Participants who continue to have a high HIV VL (≥1,000 copies/mL) after 2 months of intensive adherence counseling will be switched to second-line ART by a physician.

Participants will also be followed for a 12-month study period to assess the study outcome measures. This study will follow all aspects of South Africa's ART guidelines, except stable patients randomized to the intervention arm will receive Nurse-based care and Xpert® VL monitoring, as a comparison to the standard of care.

At the end of the 12-month study period, all participants will have a repeat CD4 count and lab-based HIV VL testing by Roche Taqman v.2.0 assay. The lab-based HIV VL testing will be important to use the same HIV VL assay to compare the primary outcomes measures. In addition, the research team will evaluate the outcome of "retention in care", which will be defined as collecting ART refills at the study exit visit.

Cost-Effectiveness Component:

The investigators will use an activity-based micro-costing approach, including time and motion studies, to estimate the costs incurred and averted, along with the primary study outcomes (viral suppression and retention in care) to estimate the cost per HIV-positive person virally suppressed and retained in care in the Intervention Group, as compared to the Standard-of-Care Group.

Time and motion studies will determine the nurse time necessary to conduct the point-of-care HIV VL testing and the clinical visit with a stable HIV-infected patient. Time and motion studies will be conducted during study initiation and again when the intervention is running at full capacity. An experienced research assistant will collect data on the time required to complete each step of the chronic care visit (VL testing, clinical assessment, counseling) for both study arms. Initial results will be shared with the teams to implement strategies for improved efficiency. Observing multiple visits will allow estimation of the average time taken for each step; the time taken for research purposes (e.g. data collection) will be noted separately from the estimated time needed for monitoring. Multiple staff will be observed to capture the range of time required for a successful real-time chronic HIV care. Interviews with study staff will also quantify the effort required for each step of visit. Through time and motion studies the number of participants who could be supported by a clinic will be estimated. The staff time taken for the intervention captures the opportunity cost of the chronic care intervention, i.e. staff time that could be spent on a different program. The micro-costing data, time and motion studies, and clinical outcomes will be used to estimate the average cost per HIV-positive client achieving viral suppression and retained in care in the chronic care model compared to the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected and receiving antiretroviral therapy (ART)
* Receiving care at Prince Cyril Zulu Clinic in Durban
* Stable on Current ART Regimen and due the 6 month follow-up visit post ART initiation
* Willing/able to provide written informed consent to participate in the stud

Exclusion Criteria:

* Have significant signs/symptoms of illness that requires active medical care by a clinic doctor.
* Does not plan to receive HIV care at the Prince Cyril Zulu Communicable Diseases Clinic for the following 12 months.
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Composite measure of virological suppression and retention in care | 12 months post enrollment
  HIV VL <200 copies/mL at 12-month study visit

SECONDARY OUTCOMES:
Proportion retained in care | 12 months post enrollment
  Proportion of patients collecting ART at the 12-month study visit
Time to detection | Every 2 months within the 12-month follow up period
  Time to detection of virological failure, subsequent intensive adherence counselling, and initiation of second line regimen
Entry into CCMDD | Every 2 months between 6 and 12 months post enrollment
  Proportion of patients entered appropriately into CCMDD, and time to appropriate entry into CCMDD
Average cost per HIV-positive client | 12 months post enrollment
  Average cost per HIV-positive client achieving viral suppression and retained in care
Number of clinical visits | 12 months post enrollment
  Mean number of clinical visits per patient
Loss to follow up or mortality | 12 months post enrollment
  Proportion lost to follow up or deceased
Change in CD4 count | 12 months post enrollment
  Mean change in CD4 count from enrolment to 12-month study exit visit
Proportion on same ART regimen | 12 months post enrollment
  Proportion of patients collecting ART at the 12-month study visit

CONTACTS AND LOCATIONS:
Overall Officials: Paul Drain, MD, MPH, Principal Investigator — University of Washington; Nigel Garrett, MBBS, MSc, Principal Investigator — Centre for the AIDS Programme of Research in South Africa (CAPRISA)
Locations (1):
- Centre for the AIDS Programme of Research in South Africa (CAPRISA), University of KwaZulu-Natal, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all outcome measures will be made available after study completion
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Dorward J, Garrett N, Quame-Amaglo J, Samsunder N, Ngobese H, Ngomane N, Moodley P, Mlisana K, Schaafsma T, Donnell D, Barnabas R, Naidoo K, Abdool Karim S, Celum C, Drain PK. Protocol for a randomised controlled implementation trial of point-of-care viral load testing and task shifting: the Simplifying HIV TREAtment and Monitoring (STREAM) study. BMJ Open. 2017 Sep 27;7(9):e017507. doi: 10.1136/bmjopen-2017-017507. PMID 28963304
- [Derived] Wang M, Violette LR, Dorward J, Ngobese H, Sookrajh Y, Bulo E, Quame-Amaglo J, Thomas KK, Garrett N, Drain PK. Delivery of Community-based Antiretroviral Therapy to Maintain Viral Suppression and Retention in Care in South Africa. J Acquir Immune Defic Syndr. 2023 Jun 1;93(2):126-133. doi: 10.1097/QAI.0000000000003176. PMID 36796353
- [Derived] Msimango L, Gibbs A, Shozi H, Ngobese H, Humphries H, Drain PK, Garrett N, Dorward J. Acceptability of point-of-care viral load testing to facilitate differentiated care: a qualitative assessment of people living with HIV and nurses in South Africa. BMC Health Serv Res. 2020 Nov 25;20(1):1081. doi: 10.1186/s12913-020-05940-w. PMID 33239012
- [Derived] Dorward J, Msimango L, Gibbs A, Shozi H, Tonkin-Crine S, Hayward G, Butler CC, Ngobese H, Drain PK, Garrett N. Understanding how community antiretroviral delivery influences engagement in HIV care: a qualitative assessment of the Centralised Chronic Medication Dispensing and Distribution programme in South Africa. BMJ Open. 2020 May 15;10(5):e035412. doi: 10.1136/bmjopen-2019-035412. PMID 32414827
- [Derived] Drain PK, Dorward J, Violette LR, Quame-Amaglo J, Thomas KK, Samsunder N, Ngobese H, Mlisana K, Moodley P, Donnell D, Barnabas RV, Naidoo K, Abdool Karim SS, Celum C, Garrett N. Point-of-care HIV viral load testing combined with task shifting to improve treatment outcomes (STREAM): findings from an open-label, non-inferiority, randomised controlled trial. Lancet HIV. 2020 Apr;7(4):e229-e237. doi: 10.1016/S2352-3018(19)30402-3. Epub 2020 Feb 24. PMID 32105625
- [Derived] Dorward J, Drain PK, Osman F, Sookrajh Y, Pillay M, Moodley P, Garrett N. Short Communication: Early Antiretroviral Therapy Is Associated with Better Viral Suppression and Less HIV Drug Resistance After Implementation of Universal Treatment in South Africa. AIDS Res Hum Retroviruses. 2020 Apr;36(4):297-299. doi: 10.1089/AID.2019.0206. Epub 2019 Dec 4. PMID 31663368
- [Derived] Dorward J, Yende-Zuma N, Samsunder N, Karim QA, Drain PK, Garrett N. Clinic-Based Evaluation of a Point-of-Care Creatinine Assay to Screen for Renal Impairment Among HIV-Positive Patients Receiving Tenofovir Disoproxil Fumarate. J Acquir Immune Defic Syndr. 2018 Apr 1;77(4):e36-e39. doi: 10.1097/QAI.0000000000001613. No abstract available. PMID 29271830